CLINICAL TRIAL: NCT04221308
Title: Evaluation of Inflammatory Markers in Single Port Laparoscopic and Vaginal Hysterectomies: A Retrospective Study in Kocaeli, Northwest Turkey
Brief Title: Inflammatory Markers in Natural Orifice Hysterectomies
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, mehmet ozsurmeli, medical doctor, Derince Training and Research Hospital
Other Study IDs: 23068423
Record Dates: First submitted 2020-01-01; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Gynecologic Disease; Inflammation
Keywords: inflammation mediators; lymphocyte activation; natural orifice endoscopic surgery; neutrophil activation; platelet activation; vaginal hysterectomy
MeSH Terms: conditions — Genital Diseases, Female; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- single port laparoscopic hysterectomies: Between 2018 and 2019, data obtained from patients in the SLH and VH groups were reviewed retrospectively. The preoperative and postoperative hematocrit (HCT), hemoglobin (HB), white blood cell (WBC), platelet (PLR), and neutrophil-lymphocyte (NLR) ratios and values were compared as well as the demographic characteristics of the patients.
  Interventions: Device: Single port laparoscopic systems
- Vaginal hysterectomies: Between 2018 and 2019, data obtained from patients in the SLH and VH groups were reviewed retrospectively. The preoperative and postoperative hematocrit (HCT), hemoglobin (HB), white blood cell (WBC), platelet (PLR), and neutrophil-lymphocyte (NLR) ratios and values were compared as well as the demographic characteristics of the patients.

INTERVENTIONS:
Device: Single port laparoscopic systems — The first assistant handles the scope from the patient's right side. The second assistant, who is positioned between the legs of the patient, inserts a uterine manipulator (Rumi System; Cooper Surgical, CT). At the beginning of the surgery, a 1.5 to 2.5 cm vertical incision is made within the umbilicus using the open Hasson approach. After the bottom retractor ring of the wound retractor component of the Octo-Port is inverted (DalimSurgNet, Seoul, Korea), it is inserted through the incision deep in the peritoneum. Carbon dioxide is insufflated through the gas valve of the Octo-Port to maintain intra-abdominal pressure at 10 to 12 mm Hg. Through the 10 mm channels of the Octo-Port, a 10 mm, 30° rigid laparoscope is introduced. Rigid laparoscopic instruments are introduced through the 5 mm channels of the Octo-Port. The utero-ovarian ligament or infundibulopelvic ligament, uterine vessels, and uterine ligaments are transected by using the 5 mm LigaSure vessel sealer device
  Groups: single port laparoscopic hysterectomies

SUMMARY:
The authors aimed to detect inflammatory marker changes in two natural orifice hysterectomies: single-port laparoscopic hysterectomy (SLH) and vaginal hysterectomy (VH).

Between 2018 and 2019, data obtained from patients in the SLH and VH groups were reviewed retrospectively. The preoperative and postoperative hematocrit (HCT), hemoglobin (HB), white blood cell (WBC), platelet (PLR), and neutrophil-lymphocyte (NLR) ratios and values were compared as well as the demographic characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* hysterectomy requirement with any conditions in gynecologic diseases

Exclusion Criteria:

* patients with a chronic disease (e.g., hypertension, diabetes mellitus, and rheumatologic, nephrological, and hematological diseases)
* the presence of active infection
* using of corticosteroid, acetylsalicylic acid, or anticoagulant
* cystocele or rectocele repair with mesh

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women without any other medical problem who need hysterectomy for any condition
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in hematocrit levels | 1 day
  Hematocrit (%) levels in the first 24 hours after single port laparoscopic or vaginal hysterectomies were compared.
Changes in hemoglobin levels | 1 day
  Hemoglobin levels in the first 24 hours after single port laparoscopic or vaginal hysterectomies were compared.
Changes in white blood cell levels | 1 day
  white blood cell (x103/mm3), in the first 24 hours after single port laparoscopic or vaginal hysterectomies were compared.
Changes in neutrophil-lymphocyte and platelet-lymphocyte ratio | 1 day
  neutrophil-lymphocyte and platelet-lymphocyte ratio in the first 24 hours after single port laparoscopic or vaginal hysterectomies were compared.

CONTACTS AND LOCATIONS:
Overall Officials: mehmet ozsurmeli, Principal Investigator — Derince Training and Research Hospital
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garry R. Health economics of hysterectomy. Best Pract Res Clin Obstet Gynaecol. 2005 Jun;19(3):451-65. doi: 10.1016/j.bpobgyn.2005.01.010. Epub 2005 Mar 2. PMID 15985258
- [Background] Yoon BS, Seong SJ, Kim IH, Song T, Kim ML, Kim MK. Operative outcomes of single-port-access laparoscopy-assisted vaginal hysterectomy compared with single-port-access total laparoscopic hysterectomy. Taiwan J Obstet Gynecol. 2014 Dec;53(4):486-9. doi: 10.1016/j.tjog.2013.07.003. PMID 25510688
- [Background] AAGL Advancing Minimally Invasive Gynecology Worldwide. AAGL position statement: route of hysterectomy to treat benign uterine disease. J Minim Invasive Gynecol. 2011 Jan-Feb;18(1):1-3. doi: 10.1016/j.jmig.2010.10.001. Epub 2010 Nov 6. No abstract available. PMID 21059487
- [Background] ACOG Committee Opinion No. 444: choosing the route of hysterectomy for benign disease. Obstet Gynecol. 2009 Nov;114(5):1156-1158. doi: 10.1097/AOG.0b013e3181c33c72. PMID 20168127
- [Background] Nieboer TE, Hendriks JC, Bongers MY, Vierhout ME, Kluivers KB. Quality of life after laparoscopic and abdominal hysterectomy: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):85-91. doi: 10.1097/AOG.0b013e31823d3b00. PMID 22183215
- [Background] Nieboer TE, Johnson N, Lethaby A, Tavender E, Curr E, Garry R, van Voorst S, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD003677. doi: 10.1002/14651858.CD003677.pub4. PMID 19588344
- [Background] Gynecol Surg. 2013; 10:117-122
- [Background] J Obstet Gynaecol. 2019; 26:1-5.
- [Background] Cruickshank AM, Fraser WD, Burns HJ, Van Damme J, Shenkin A. Response of serum interleukin-6 in patients undergoing elective surgery of varying severity. Clin Sci (Lond). 1990 Aug;79(2):161-5. doi: 10.1042/cs0790161. PMID 2167805
- [Background] Allendorf JD, Bessler M, Whelan RL, Trokel M, Laird DA, Terry MB, Treat MR. Postoperative immune function varies inversely with the degree of surgical trauma in a murine model. Surg Endosc. 1997 May;11(5):427-30. doi: 10.1007/s004649900383. PMID 9153168
- [Background] Lennard TW, Shenton BK, Borzotta A, Donnelly PK, White M, Gerrie LM, Proud G, Taylor RM. The influence of surgical operations on components of the human immune system. Br J Surg. 1985 Oct;72(10):771-6. doi: 10.1002/bjs.1800721002. PMID 2412626
- [Background] Iwase M, Kondo G, Watanabe H, Takaoka S, Uchida M, Ohashi M, Nagumo M. Regulation of Fas-mediated apoptosis in neutrophils after surgery-induced acute inflammation. J Surg Res. 2006 Jul;134(1):114-23. doi: 10.1016/j.jss.2005.10.013. Epub 2005 Dec 27. PMID 16376940
- [Background] Ogawa K, Hirai M, Katsube T, Murayama M, Hamaguchi K, Shimakawa T, Naritake Y, Hosokawa T, Kajiwara T. Suppression of cellular immunity by surgical stress. Surgery. 2000 Mar;127(3):329-36. doi: 10.1067/msy.2000.103498. PMID 10715990
- [Background] Collet D, Vitale GC, Reynolds M, Klar E, Cheadle WG. Peritoneal host defenses are less impaired by laparoscopy than by open operation. Surg Endosc. 1995 Oct;9(10):1059-64. doi: 10.1007/BF00188987. PMID 8553203
- [Background] Sietses C, Wiezer MJ, Eijsbouts QA, van Leeuwen PA, Beelen RH, Meijer S, Cuesta MA. The influence of laparoscopic surgery on postoperative polymorphonuclear leukocyte function. Surg Endosc. 2000 Sep;14(9):812-6. doi: 10.1007/s004640010080. PMID 11000359
- [Background] Malik E, Buchweitz O, Muller-Steinhardt M, Kressin P, Meyhofer-Malik A, Diedrich K. Prospective evaluation of the systemic immune response following abdominal, vaginal, and laparoscopically assisted vaginal hysterectomy. Surg Endosc. 2001 May;15(5):463-6. doi: 10.1007/s004640000348. Epub 2001 Mar 13. PMID 11353962
- [Background] Choi YS, Shin KS, Choi J, Park JN, Oh YS, Rhee TE. Single-port access laparoscopy-assisted vaginal hysterectomy: our initial experiences with 100 cases. Minim Invasive Surg. 2012;2012:543627. doi: 10.1155/2012/543627. Epub 2012 Sep 4. PMID 22988497
- [Background] Liliana M, Alessandro P, Giada C, Luca M. Single-port access laparoscopic hysterectomy: a new dimension of minimally invasive surgery. J Gynecol Endosc Surg. 2011 Jan;2(1):11-7. doi: 10.4103/0974-1216.85273. PMID 22442528
- [Background] Romanelli JR, Earle DB. Single-port laparoscopic surgery: an overview. Surg Endosc. 2009 Jul;23(7):1419-27. doi: 10.1007/s00464-009-0463-x. Epub 2009 Apr 4. No abstract available. PMID 19347400
- [Background] Gynecol Surg. 2010; 7(2):143-148
- [Background] Lee YY, Kim TJ, Kim CJ, Kang H, Choi CH, Lee JW, Kim BG, Lee JH, Bae DS. Single-port access laparoscopic-assisted vaginal hysterectomy: a novel method with a wound retractor and a glove. J Minim Invasive Gynecol. 2009 Jul-Aug;16(4):450-3. doi: 10.1016/j.jmig.2009.03.022. Epub 2009 May 31. PMID 19487164
- [Background] Terzi H, Biler A, Turkay U, Kale A. A comparison of novel laparoscopic suturing techniques in single-port surgery. Minim Invasive Ther Allied Technol. 2019 Dec;28(6):338-343. doi: 10.1080/13645706.2019.1567554. Epub 2019 Feb 22. PMID 30793638
- [Background] Goolab BD. Vaginal hysterectomy and relative merits over abdominal and laparoscopically assisted hysterectomy. Best Pract Res Clin Obstet Gynaecol. 2013 Jun;27(3):393-413. doi: 10.1016/j.bpobgyn.2013.01.003. Epub 2013 Apr 18. PMID 23602203
- [Background] Dedden SJ, Geomini PMAJ, Huirne JAF, Bongers MY. Vaginal and Laparoscopic hysterectomy as an outpatient procedure: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2017 Sep;216:212-223. doi: 10.1016/j.ejogrb.2017.07.015. Epub 2017 Jul 22. PMID 28810192
- [Background] Fornara P, Doehn C, Seyfarth M, Jocham D. Why is urological laparoscopy minimally invasive? Eur Urol. 2000 Mar;37(3):241-50. doi: 10.1159/000052351. PMID 10720847
- [Background] Slade MS, Simmons RL, Yunis E, Greenberg LJ. Immunodepression after major surgery in normal patients. Surgery. 1975 Sep;78(3):363-72. PMID 1098195
- [Background] Sietses C, Wiezer MJ, Eijsbouts QA, Beelen RH, van Leeuwen PA, von Blomberg BM, Meijer S, Cuesta MA. A prospective randomized study of the systemic immune response after laparoscopic and conventional Nissen fundoplication. Surgery. 1999 Jul;126(1):5-9. doi: 10.1067/msy.1999.98702. PMID 10418585
- [Background] Gupta A, Watson DI. Effect of laparoscopy on immune function. Br J Surg. 2001 Oct;88(10):1296-306. doi: 10.1046/j.0007-1323.2001.01860.x. PMID 11578282
- [Background] Grace PA, Quereshi A, Coleman J, Keane R, McEntee G, Broe P, Osborne H, Bouchier-Hayes D. Reduced postoperative hospitalization after laparoscopic cholecystectomy. Br J Surg. 1991 Feb;78(2):160-2. doi: 10.1002/bjs.1800780209. PMID 1826624
- [Background] Faist E, Kupper TS, Baker CC, Chaudry IH, Dwyer J, Baue AE. Depression of cellular immunity after major injury. Its association with posttraumatic complications and its reversal with immunomodulation. Arch Surg. 1986 Sep;121(9):1000-5. doi: 10.1001/archsurg.1986.01400090026004. PMID 3741094
- [Background] Sandberg EM, la Chapelle CF, van den Tweel MM, Schoones JW, Jansen FW. Laparoendoscopic single-site surgery versus conventional laparoscopy for hysterectomy: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 May;295(5):1089-1103. doi: 10.1007/s00404-017-4323-y. Epub 2017 Mar 29. PMID 28357561
- [Background] Ramirez PT. Single-port laparoscopic surgery: is a single incision the next frontier in minimally invasive gynecologic surgery? Gynecol Oncol. 2009 Aug;114(2):143-4. doi: 10.1016/j.ygyno.2009.06.007. No abstract available. PMID 19559942
- [Background] Fader AN, Escobar PF. Laparoendoscopic single-site surgery (LESS) in gynecologic oncology: technique and initial report. Gynecol Oncol. 2009 Aug;114(2):157-61. doi: 10.1016/j.ygyno.2009.05.020. Epub 2009 May 28. PMID 19481243